CLINICAL TRIAL: NCT04845451
Title: The Presence and Role of Zygomatic-temporal Neuroma Triggering Cluster Headache: Resection of a Neuroma in the Long-term Resolution of Trigeminal Cluster Symptoms
Brief Title: The Presence and Role of Zygomatic-temporal Neuroma Triggering Cluster Headache
Status: Completed | Type: Observational
Sponsor: FARO T. OWIESY, M.D (Other)
Collaborators: Ohsi, Steven, M.D (Unknown); Radfar, Amir, M.D (Unknown)
Responsible Party: Sponsor-Investigator, FARO T. OWIESY, M.D, principal investigator, Corona Doctors Medical Clinics, Inc.
Organization: Corona Doctors Medical Clinics, Inc. (Other)
Other Study IDs: CoronaDMC
Record Dates: First submitted 2021-04-10; First posted 2021-04-15 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Cluster Headache; Craniofacial Pain Syndrome
Keywords: cluster headache; neuralgic headache
MeSH Terms: conditions — Cluster Headache; Facial Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Minimal surgical exploration for a neuroma — Orientation marking of the trigger point by injectable sterile methylene blue dye 0.1ml. Marking a 2-3-centimeter long incision line 7 mm from the Neuroma marking on the skin. Local anesthesia using plain 2% lidocaine infiltration of the circumferential exploratory area. Sterile prep and drape in surgical fashion. Meticulous exploratory preparation of the subcutaneous tissue 20 mm at each side of the incision line. Appropriate visibility of the ZT nerve branches embedded in lipomatous and connective tissue over the temporal fascia. Exploratory visualization of the subcutaneous marked tissue by methylene blue using a binocular magnification eases visualization. Using an Adson tissue forceps with side grasping teeth, now an exploratory touch of the above and distal of the marking would deliver the hypersensitive painful Neuroma tissue for sharp excision using surgical scissors. Control of bleeding and skin closure. Sterile pressure dressing. Specimen be sent to pathologic examination.
  Other Names: Clusterotomy

SUMMARY:
Role of a neuroma of zygomatic-temporal in triggering of a cluster headache. Exploratory diagnosis, resection, and pathological examination of tumor anticipated

.

DETAILED DESCRIPTION:
An anatomical coordinated communication of a Cluster Circuit turned on by Zygomatico-Temporal neuroma, a malicious possibly nontraumatic, neoplastic tissue coding and decoding itself upon autonomic release of neurotransmitter(s). Exhaustion of neurotransmitter synthesis turns out the explosions of pain-symptoms off.

Poor attention to the characterization of a peripheral neuroma of trigeminal nerve branch deranged attention to central(CNS) characterization of Cluster Symptoms.

This study based on our experimental results of minimal surgical procedure to explore, diagnose and resect a Zygomatico-Temporal neuroma in the temple of patients suffering from EpisodicChronic, Cluster Headache-ECCH. The goal is to light on this speculation in a novel analysis of events to put an end to devastating catastrophic headaches. Detailed anatomical components loci of the autonomic symptoms in the cluster headache reveal the presence of an electrical neural circuit.

The extracranial circuit components of ECCH reflects the anatomical nerve components participating reflection of the single circumscribed symptom:

1. Zygomatico-Temporal-neuroma
2. Zygomatic nerve V-II
3. Intraorbital communicants rami
4. Lacrimal nerve V-I
5. Ophthalmic nerve Intraorbital routing, supraorbital nerves, the upper eyelid, the conjunctiva and cornea of the eye, the nose (including the tip of the nose, except alae nasi), the nasal mucosa, the frontal sinuses. V-I
6. Optic nerve via ophthalmic nerve routing and electricity propagation.
7. Pterygopalatine ganglion as peripheral and CNS coordinator center.

An intracranial CNS reaction follows in response to the perception of pain materialized in neuroimaging during the activity of ECCH.

ELIGIBILITY:
Inclusion Criteria:

- Cluster headache

Exclusion Criteria:

* Malignant hypertension,
* Brain tumors,
* Cerebral vascular abnormalities,
* Presence of a brain or nerve electro stimulator.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ٠patients suffering from episodic and chronic cluster headaches
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Presence of Neuroma | 6 months
  Zygomaticotemporal neuroma as trigger of Episodic and Chronic Cluster headache
Resolution of Cluster Headache attacks | 6 months
  Resection of a ZT-neuroma may eradicate Cluster Headache trigger

CONTACTS AND LOCATIONS:
Overall Officials: Faro T Owiesy, M.D., Principal Investigator — CORONA DOCTORS MEDICAL CLINICS; Steven Ohsie, M.D, Study Chair — Affiliated Patholgy; Amir Radfar, M.D,MPH, Study Director — Corona doctors medical clinics
Locations (1):
- Corona Doctors Medical Clinics Inc, Corona, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Presentation by poster, article, and on-demand providing the data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6-9 months
Access Criteria: scientific, clinicians, national and international sources. No limitations